CLINICAL TRIAL: NCT07339501
Title: Cystic Artery Preservation : an Additional Step for Safe Laparoscopic Cholecystectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Suez University (Other)
Collaborators: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmad Ali Maklad, lecturer of general surgery, Suez University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SVU MED SUR011
Record Dates: First submitted 2025-11-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Chronic Calculous Cholecystitis
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) (Active Comparator)
  Interventions: Procedure: The patients will be operated on for laparoscopic cholecystectomy with preservation of cystic artery a
- group B (Placebo Comparator)
  Interventions: Procedure: The patients will be operated on for laparoscopic cholecystectomy with clipping or cauterization of cystic artery

INTERVENTIONS:
Procedure: The patients will be operated on for laparoscopic cholecystectomy with preservation of cystic artery a — The patients will be operated on for laparoscopic cholecystectomy with preservation of cystic artery for save cholecystectomy
  Arms: group (A)
Procedure: The patients will be operated on for laparoscopic cholecystectomy with clipping or cauterization of cystic artery — The patients will be operated on for laparoscopic cholecystectomy with clipping or cauterization of cystic artery
  Arms: group B

SUMMARY:
Our aim is to feature additional steps for safe cholecystectomy by preserving the cystic artery.

ELIGIBILITY:
Inclusion Criteria:

* 1-Patients with symptomatic gall bladder stones. 2-Patients with normal coagulation profile.

Exclusion Criteria:

* 1- Patients with hepatic co-morbidity especially (cirrhosis). 2-Patients with previous upper abdominal surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Patients will be followed up by Abdominal ultrasound for post operative abdominal collection | one month
  Follow up with ultrasound to evaluate if there's bleeding or not after preserving the cystic artery

CONTACTS AND LOCATIONS:
Locations (1):
- Suez University, Suez, Egypt

IPD SHARING:
Plan to Share IPD: Undecided